CLINICAL TRIAL: NCT03090334
Title: A B-D-Glucan Driven Antifungal Stewardship Approach to Manage Empirical Therapy in Patients at Very High Risk for Invasive Candidiasis: a Randomized Controlled Trial
Brief Title: A B-D-Glucan Driven Antifungal Stewardship Approach for Invasive Candidiasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient rate of accrual due to the start of a concomitant similar study
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Maddalena Giannella, MD, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BDG-ETHIC
Record Dates: First submitted 2017-03-18; First posted 2017-03-24 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Invasive Candidiases; Abdominal Infection
Keywords: beta-d-glucan; abdominal candidiasis
MeSH Terms: conditions — Candidiasis, Invasive; Intraabdominal Infections

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Care provider will be blinded to result of BG in patients enrolled in the standard of care arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- De-escalation (Experimental): In this group, investigators will manage the antifungal therapy according to the BG levels as follows:
  1. antifungal therapy will be stopped immediately after the BG response in case of serum BG <80 pg/ml in presence of clinical stability (CS);
  2. antifungal therapy will be continued until further BG determination, both for BG levels between 80-200 pg/ml and for BG <80 pg/ml in patients without CS. In these cases, if the following BG value is <80 pg/ml antifungal therapy will be stopped independently from the CS achievement.
  3. antifungal therapy will be continued until day 10 for BG levels >200 pg/ml
  Interventions: Diagnostic Test: De-escalation
- Standard of care (No Intervention): In this group antifungal treatment will be continued until clinician's decision.
  Investigators will be blinded to the BG levels of patients enrolled in this arm, The BG results will be faxed directly to the coordinating center.

INTERVENTIONS:
Diagnostic Test: De-escalation — Antifungal therapy will be stopped according with BG results
  Arms: De-escalation

SUMMARY:
This is a multicenter, prospective, open-label, randomized trial. Patients with severe abdominal condition developing severe sepsis or septic shock and receiving broad spectrum antibiotic and antifungal treatment will be randomized (1:1) to:

1. discontinue antifungal treatment based on negative (<80 pg/ml) result of 1,3 beta-d-glucan performed on day 0,3,6 and 10
2. continue antifungal treatment according with attending physician's decision.

DETAILED DESCRIPTION:
Primary objective:

Our objective is to establish whether a strategy based on beta-d-glucan (BG) assessment could achieve reduced antifungal consumption in patients with severe abdominal condition developing severe sepsis and septic shock without any impact on the outcome Secondary objectives i) Assess the accuracy of BG in the diagnosis of invasive candidiasis (IC) in in critically ill patients with a severe abdominal condition who develop severe sepsis or septic shock.

ii) Describe the changes over the time of BG value according with colonization status, infection or none the aforementioned events.

Material and Methods Study design: a multicenter, open label, randomized trial Population: all the patients with a severe abdominal condition who develop a severe sepsis or septic shock.

1. Inclusion Criteria:

   1. adult (≥ 18 year) patients;
   2. signed informed consent before surgical procedure;
   3. severe sepsis or septic shock;
   4. at least one of the following conditions: i) post-operative peritonitis, ii) recurrent gastrointestinal perforation, iii) post-operative hepatobiliary and/or pancreatic disorders including necrotizing pancreatitis, iv) post-operative intra-abdominal abscess, and v) anastomotic leak.
2. Exclusion criteria a. diagnosis of candidiasis before the enrollment b. exposure in the past 30 days to any antifungal treatment or diagnosis of invasive fungal infection; c. pregnancy or lactation; d. history of allergy to any of the antifungal drugs; e. major immunosuppression conditions including: i. neutropenia (<0.5 × 109 neutrophils/L [<500 neutrophils/mm3] for >10 days), ii. receipt of an allogeneic stem cell transplant or solid organ transplantation, iii. inherited severe immunodeficiency (such as chronic granulomatous disease or severe combined immunodeficiency), iv. HIV infection with lymphocyte T CD4+ cell count < 200/mmc. f. patients with poor prognosis or unable to sign informed consent.

Procedures Pre-randomization procedures

At the time of patient enrollment (within 24 h from onset of severe sepsis/septic shock), a standardized diagnostic work-up must be performed including at least:

i) two sets of blood cultures; ii) 5 surveillance cultures (rectal swab, urine culture, pharyngeal swab, axillary swab, groin swab).

iii) in case of re-intervention or percutaneous drainage: Gram stain and culture of intra-abdominal samples; iv) serum BG determination. Antibiotic and antifungal empirical therapy should be started immediately after collection of microbiological samples according with a predefined standard of care (see appendix 1). Once completed this procedures patients will proceed to randomization.

Randomization Patient eligible for the study after the beginning of antifungal therapy will be randomized 1:1 to receive (Group A) a BG driven de-escalation strategy or (Group B) a course of antifungal treatment based on the care provider's decision.

In both groups, if cultures yield invasive candidiasis (see below) the patient will be managed in according with guidelines and excluded from the per-protocol analysis.

In both groups, BG determination will be repeated at day +3, +6 and +10 after starting antifungal therapy.

Randomization will be carried out providing closed envelopes to the participating centers immediately before the study onset.

ELIGIBILITY:
Inclusion Criteria:

* a. adult (≥ 18 year) patients; b. signed informed consent before surgical procedure; c. severe sepsis or septic shock; d. at least one of the following conditions: i) post-operative peritonitis, ii) recurrent gastrointestinal perforation, iii) post-operative hepatobiliary and/or pancreatic disorders including necrotizing pancreatitis, iv) post-operative intra-abdominal abscess, and v) anastomotic leak.

Exclusion Criteria:

* a. diagnosis of candidiasis before the enrollment b. exposure in the past 30 days to any antifungal treatment or diagnosis of invasive fungal infection; c. pregnancy or lactation; d. history of allergy to any of the antifungal drugs; e. major immunosuppression conditions including: i. neutropenia (<0.5 × 109 neutrophils/L [<500 neutrophils/mm3] for >10 days), ii. receipt of an allogeneic stem cell transplant or solid organ transplantation, iii. inherited severe immunodeficiency (such as chronic granulomatous disease or severe combined immunodeficiency), iv. HIV infection with lymphocyte T CD4+ cell count < 200/mmc. f. patients with poor prognosis or unable to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Antifungal consumption | 28 days
  Days of antifungal consumption will be compared between the two groups
Mortality | 28 days
  28-day mortality will be compared between the two groups
Length of stay | 28 days
  Length of stay in ICU will be compared between the two groups

SECONDARY OUTCOMES:
Accuracy of BG | 28 days
  sensitivity, specificity, positive predictive value, negative predictive value of BG in the diagnosis of invasive candidiasis

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospealiero Universitaria di Bologna Policlinico S.Orsola-Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bassetti M, Marchetti M, Chakrabarti A, Colizza S, Garnacho-Montero J, Kett DH, Munoz P, Cristini F, Andoniadou A, Viale P, Rocca GD, Roilides E, Sganga G, Walsh TJ, Tascini C, Tumbarello M, Menichetti F, Righi E, Eckmann C, Viscoli C, Shorr AF, Leroy O, Petrikos G, De Rosa FG. A research agenda on the management of intra-abdominal candidiasis: results from a consensus of multinational experts. Intensive Care Med. 2013 Dec;39(12):2092-106. doi: 10.1007/s00134-013-3109-3. Epub 2013 Oct 9. PMID 24105327
- [Background] Kollef M, Micek S, Hampton N, Doherty JA, Kumar A. Septic shock attributed to Candida infection: importance of empiric therapy and source control. Clin Infect Dis. 2012 Jun;54(12):1739-46. doi: 10.1093/cid/cis305. Epub 2012 Mar 15. PMID 22423135
- [Background] Maubon D, Garnaud C, Calandra T, Sanglard D, Cornet M. Resistance of Candida spp. to antifungal drugs in the ICU: where are we now? Intensive Care Med. 2014 Sep;40(9):1241-55. doi: 10.1007/s00134-014-3404-7. Epub 2014 Aug 5. PMID 25091787
- [Background] Clancy CJ, Nguyen MH. Finding the "missing 50%" of invasive candidiasis: how nonculture diagnostics will improve understanding of disease spectrum and transform patient care. Clin Infect Dis. 2013 May;56(9):1284-92. doi: 10.1093/cid/cit006. Epub 2013 Jan 11. PMID 23315320